CLINICAL TRIAL: NCT02997124
Title: Transversus Abdominis Plane Block Supplementation During Iliac Crest Bone Graft Harvest - Its Influence on Postoperative Parameters
Brief Title: Transversus Abdominis Plane Block in Iliac Crest harvest-is it Beneficial?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Vigil Peter, Assistant Professor, Department of Anesthesia, Jubilee Mission Medical College and Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07/16/IEC/JMMC&RI
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Pain, Postoperative
Keywords: Alveolar bone grafting; delirium; early ambulation
MeSH Terms: conditions — Pain, Postoperative; Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local Infiltration with TAP block (Experimental): Ultrasound guided Transversus Abdominis Plane block is administered intraoperatively using 0.2% Ropivacaine.
  Interventions: Procedure: local infiltration and TAP block
- Local Infiltration only (Experimental): Local Infiltration with 0.2% Ropivacaine.
  Interventions: Procedure: local infiltration only

INTERVENTIONS:
Procedure: local infiltration and TAP block — Local infiltration of the iliac crest harvest site along with TAP block using 0.2 % Ropivacaine is done
  Arms: Local Infiltration with TAP block
Procedure: local infiltration only — Only local infiltration with 0.2% Ropivacaine of the iliac crest harvest site is done.
  Arms: Local Infiltration only

SUMMARY:
The purpose of this study is to determine whether a supplemental Transversus Abdominis Plane block administered intraoperatively improves the postoperative parameters in patients undergoing Alveolar bone grafting with iliac crest harvest. It also aims to find out if there is a decrease in the incidence of chronic pain or numbness at the harvest site.

DETAILED DESCRIPTION:
This study is a prospective, randomised, parallel group, single - centre trial evaluating the postoperative parameters in patients receiving supplemental Transversus Abdominis Plane block for anterior iliac crest harvest. It was conducted in 143 patients undergoing Alveolar bone grafting with iliac crest bone graft.

Methodology:

Informed consent and approval of local ethics and research committee in Jubilee Mission Medical College and Research Institute, Thrissur, India was obtained prior to initiation of the study. A pilot study was done to determine the efficacy of the additional TAP block. The results showed that the intervention improved patient analgesia and reduced the requirement for rescue analgesics. A minimum sample size of 65 patients was calculated for each group to obtain a power of 80% and confidence interval of 95%. 143 patients aged between 7 and 22 years posted for Alveolar bone grafting with anterior iliac crest harvest were assessed in the study. Only those undergoing Alveolar bone grafting as a part of the reconstructive procedure for cleft lip and palate were considered for the study. The patients who had difficulty in mentation and communication,bleeding disorders, hepatic problems, infection of the abdominal wall, renal dysfunction as well as allergy to the local anaesthetic were excluded from the study. Patients undergoing revision surgeries were also excluded from the study. All the candidates were randomly alloted to either of the two groups, using a computer - generated number.

All the patients were premedicated with Midazolam 0.15mg kg-1 and Glycopyrolate 0.01mg kg-1 Anaesthesia was induced with Propofol 2 mg kg -1 and Fentanyl 2 mcg kg-1 .Vecuronium 0.1 mg kg-1 was given to facilitate orotracheal intubation with a cuffed tube.Anaesthesia was maintained with oxygen, nitrous oxide and sevoflurane. Prior to incision, all the patients were given wound infiltration with 0.75 ml kg-1 of 0.2% Ropivacaine at the graft harvest site. Those in group A received an additional ultrasound guided Transversus Abdominis Plane block with a similar volume and concentration of Ropivacaine.

At the end of the surgical procedure, the patients were extubated awake, after giving I / V Neostigmine 0.05 mg kg-1. Just prior to extubation, I/V Tramadol 0.5 mg kg-1 was given for the pain in the postoperative period. In the recovery room, the pain and emergence delirium were assessed by an independent observer every ten minutes during the first postoperative hour.These were evaluated using the FLACC Behavioural Pain Assessment Scale and WATCHA Scale respectively. They were subsequently shifted to the postoperative ward.

The next time point of assessment was 24 hours post - surgery, when the patient's pain and ambulatory status were evaluated. The pain was ranked using the five - point verbal ranking score. It was ranked as no pain, light pain, moderate pain, severe pain and intolerable pain, with a score of 0,1,2,3 and 4 respectively. The total number of rescue analgesics demanded by the patient on the first postoperative day was noted.Ambulatory status was graded using one - day Cumulated Ambulatory Score.

The patients were followed up and questioned at six weeks and twelve weeks post operatively for the presence of chronic pain, numbness or wound healing problems at the harvest site.

ELIGIBILITY:
Inclusion Criteria:

* Must undergo alveolar bone grafting as a part of the reconstructive procedure for cleft lip and palate

Exclusion Criteria:

* Revision procedure
* History of difficulty in mentation and communication
* Bleeding disorders, hepatic problems or renal dysfunction
* Allergy to local anaesthetic
* Presence of infection of anterior abdominal wall

Ages: 4 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 143 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mean pain scores | First hour after extubation
  Mean pain scores were assessed using the FLACC Behavioural Pain Assessment Scale,
Emergence delirium | First hour after extubation
  Emergence delirium was assessed using WATCHA Scale during the first hour after extubation
Pain scores | 24 hours after surgery
  Pain scores using the five - point verbal ranking score 24 hours after surgery
Ambulatory status | 24 hours after surgery
  Ambulatory status was assessed using one - day Cumulated Ambulatory Score 24 hours after surgery

SECONDARY OUTCOMES:
Infection and delayed healing at the graft harvest site | 6 weeks after surgery
  All patients were interviewed for the presence of infection or delayed healing at the graft harvest site 6 weeks after surgery.
Chronic pain, numbness or discomfort at graft harvest site | 12 weeks after the surgery
  All the patients were reviewed 12 weeks after surgery for the presence of chronic pain, numbness or discomfort at iliac crest harvest

CONTACTS AND LOCATIONS:
Overall Officials: Vigil Peter, MD, Principal Investigator — Jubilee Mission Medical College and Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiono J, Bernard N, Bringuier S, Biboulet P, Choquet O, Morau D, Capdevila X. The ultrasound-guided transversus abdominis plane block for anterior iliac crest bone graft postoperative pain relief: a prospective descriptive study. Reg Anesth Pain Med. 2010 Nov-Dec;35(6):520-4. doi: 10.1097/AAP.0b013e3181fa117a. PMID 20975466
- [Background] Sandhu HS, Grewal HS, Parvataneni H. Bone grafting for spinal fusion. Orthop Clin North Am. 1999 Oct;30(4):685-98. doi: 10.1016/s0030-5898(05)70120-6. PMID 10471772
- [Background] Heary RF, Schlenk RP, Sacchieri TA, Barone D, Brotea C. Persistent iliac crest donor site pain: independent outcome assessment. Neurosurgery. 2002 Mar;50(3):510-6; discussion 516-7. doi: 10.1097/00006123-200203000-00015. PMID 11841718
- [Background] DeOrio JK, Farber DC. Morbidity associated with anterior iliac crest bone grafting in foot and ankle surgery. Foot Ankle Int. 2005 Feb;26(2):147-51. doi: 10.1177/107110070502600206. PMID 15737257
- [Background] Silber JS, Anderson DG, Daffner SD, Brislin BT, Leland JM, Hilibrand AS, Vaccaro AR, Albert TJ. Donor site morbidity after anterior iliac crest bone harvest for single-level anterior cervical discectomy and fusion. Spine (Phila Pa 1976). 2003 Jan 15;28(2):134-9. doi: 10.1097/00007632-200301150-00008. PMID 12544929
- [Background] Kim DH, Rhim R, Li L, Martha J, Swaim BH, Banco RJ, Jenis LG, Tromanhauser SG. Prospective study of iliac crest bone graft harvest site pain and morbidity. Spine J. 2009 Nov;9(11):886-92. doi: 10.1016/j.spinee.2009.05.006. Epub 2009 Jun 18. PMID 19540168
- [Background] O'Donnell BD, McDonnell JG, McShane AJ. The transversus abdominis plane (TAP) block in open retropubic prostatectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):91. doi: 10.1016/j.rapm.2005.10.006. No abstract available. PMID 16418039
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Kessler P, Thorwarth M, Bloch-Birkholz A, Nkenke E, Neukam FW. Harvesting of bone from the iliac crest--comparison of the anterior and posterior sites. Br J Oral Maxillofac Surg. 2005 Feb;43(1):51-6. doi: 10.1016/j.bjoms.2004.08.026. PMID 15620775
- [Background] Zijderveld SA, ten Bruggenkate CM, van Den Bergh JP, Schulten EA. Fractures of the iliac crest after split-thickness bone grafting for preprosthetic surgery: report of 3 cases and review of the literature. J Oral Maxillofac Surg. 2004 Jul;62(7):781-6. doi: 10.1016/j.joms.2003.12.018. PMID 15218554
- [Background] Rawashdeh MA, Telfah H. Secondary alveolar bone grafting: the dilemma of donor site selection and morbidity. Br J Oral Maxillofac Surg. 2008 Dec;46(8):665-70. doi: 10.1016/j.bjoms.2008.07.184. Epub 2008 Aug 29. PMID 18760515
- [Background] Kalk WW, Raghoebar GM, Jansma J, Boering G. Morbidity from iliac crest bone harvesting. J Oral Maxillofac Surg. 1996 Dec;54(12):1424-9; discussion 1430. doi: 10.1016/s0278-2391(96)90257-8. PMID 8957121